CLINICAL TRIAL: NCT02599116
Title: A Cohort Study of the Gastrointestinal Microbiome in Appendiceal Cancer With Peritoneal Spread
Brief Title: Gastrointestinal Microbiome Study of Appendiceal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercy Medical Center (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Armando Sardi, Chief Surgical Oncology at Mercy, Mercy Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MMC 2015-53
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Pseudomyxoma Peritonei; Appendiceal Neoplasm; Cancer, Appendiceal
Keywords: cytoreductive surgery; hyperthermic intraperitoneal chemotherapy; microbiome
MeSH Terms: conditions — Pseudomyxoma Peritonei; Appendiceal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microbiome cohort (Other): 1. Pre-operative (baseline) bio-specimen collection (fecal sample) and completion of two food and lifestyle questionnaires.
  2. Six to twelve weeks following cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CRS/HIPEC), post-operative bio-specimen collection (fecal sample) and completion of two food and lifestyle questionnaires
  3. Six to twelve months following cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CRS/HIPEC), post-operative bio-specimen collection (fecal sample) and completion of two food and lifestyle questionnaires
  Interventions: Other: Bio-specimen collection; Other: Questionnaire

INTERVENTIONS:
Other: Bio-specimen collection — Collection of bio-specimens (fecal sample) at 3 different time points One pre-operative collection, Two post-operative collections
Other: Questionnaire — Completion of lifestyle and food questionnaires (2) at each bio-specimen collection timepoint

SUMMARY:
This study analyzes the gastrointestinal microbiome of appendiceal cancer patients with peritoneal spread scheduled to undergo cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CRS/HIPEC). Participants will provide fecal samples pre- and post-operatively.

DETAILED DESCRIPTION:
Analysis of the human microbiome is an attempt to define how changes in the human microbiome are associated with health or disease.

Eligible participants scheduled to undergo cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CRS/HIPEC) for appendiceal cancer will provide fecal samples pre- and post-operatively. Investigators will analyze potential changes in the gastrointestinal microbiome and make comparisons to an age-matched healthy sample.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of appendiceal cancer with peritoneal spread
* Candidate for cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CRS/HIPEC)
* ≥18 and ≤ 80 years of age
* Eastern Cooperative Oncology Group performance status score of ≤2/Karnofsky performance status (KPS) ≥70%
* Signed Institutional Review Board approved informed consent

Exclusion Criteria:

* <18 years of age
* Pregnant women
* Concurrent severe medical problems unrelated to malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-12; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Determine whether the intestinal microbiome of patients with appendiceal tumors with peritoneal carcinomatosis differs from that of a healthy, age-matched cohort | 36 months
  Appendiceal cohort to healthy age-matched cohort

SECONDARY OUTCOMES:
Compare the gut microbiome of appendiceal tumors by histopathology | 36 months
  Low-grade and high-grade tumors

OTHER OUTCOMES:
Identify potential biomarkers associated with appendiceal tumors | 36 months
  Molecular profile
Identify alterations in the gut microbiome post-CRS/HIPEC | 36 months
  Compare pre-HIPEC and post-HIPEC samples

CONTACTS AND LOCATIONS:
Overall Officials: Armando Sardi, MD, Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gilbreath JJ, Semino-Mora C, Friedline CJ, Liu H, Bodi KL, McAvoy TJ, Francis J, Nieroda C, Sardi A, Dubois A, Lazinski DW, Camilli A, Testerman TL, Merrell DS. A core microbiome associated with the peritoneal tumors of pseudomyxoma peritonei. Orphanet J Rare Dis. 2013 Jul 12;8:105. doi: 10.1186/1750-1172-8-105. PMID 23844722
- See also: The American Gut Project is an open-source project to understand the microbial diversity of the human gut. — http://americangut.org/